#### RESEARCH INFORMATION SHEET

Dear. Mrs / Miss

We hereby explain that LACK OF VITAMIN D can cause bone loss and aggravate lung disease. For this reason, we will conduct research to find out whether by providing supplementation with vitamin D 1000 IU per day and Vitamin A 6000 IU / day along with lifestyle changes, mothers / sisters so that later they can increase levels of vitamin D and calcium. If the mother / sister is willing to take part in this research, then:

- 1. Interview about: age, habit of taking supplements, sun exposure and daily physical activity.
- 2. Interview about food and beverages by interviewing eating habits at each meeting.
- 3. Check your weight, height and waist circumference.
- 4. Blood draws that are carried out once, namely the present meeting of approximately 5 (five) mL for each of the tests of vitamins D and A

As a result of the blood draw, you may feel some discomfort or pain, but this can be minimized by taking blood by trained personnel and using a small syringe. The participation of mothers / sisters in this research is voluntary and mothers / sisters can refuse or resign during the research process. The advantage for mothers / sisters when participating in this research is that mothers / sisters can know their respective genetic conditions so that the appropriate type of food can be determined so that diabetes can be prevented. All data in this study are confidential.

If the mother / sister is willing to participate in this research, we will ask for her willingness to be able to sign a letter of consent to be a research participant:

# LIFESTYLE CHANGE MODELS ON TUBERCULOSIS PATIENTS: VITAMIN D AND A STUDY

The things that are not clear in this study can be asked directly, via sms or by telephone to the person in charge of this research, namely Dr. dr. Dina Keumala Sari, MG, SpGK, home address: road ring road, komp. Tasbih 2, block 5. Number 126, Medan, North Sumatra, Indonesia, telephone: 061-4256-4286, cell phone: 081397177693.

We thank you for the willingness of Mrs/Miss.

## **Informed Consent**

## LEMBAGA PENELITIAN UNIVERSITAS SUMATERA UTARA

#### LETTER OF AGREEMENT TO BE A RESEARCH PARTICIPANT

| i, the undersigned below | • | |
|---|---|---|
| Name | : | |
| Age / date of birth | : | |
| Tribe (follow your father's tr | ibal line) : | |
| Marital status | : O married O s | ingle |
| Address | : | |
| After receiving sufficient in | formation and und | erstanding the benefits of the research below |
| which is entitled: | | |
| | | NGE MODELS ON<br>5: VITAMIN D AND A STUDY |
| Voluntarily agreeing to be | included in the abo | ove research provided that at any time you are |
| harmed in any form has the | right to cancel this | agreement. |
| | | Medan,2019 |
| Who responsible for resear | ch: | Who approved |
| Dr. dr. Dina Keumala Sari N | MG, SpGK | () |
| The Witness: | | |
| ( | ) | |